CLINICAL TRIAL: NCT06095635
Title: Acute Influence of Resveratrol Supplementation and Beet Extract in Recovery After Exercise Submaximal Aerobic in Coronary Paths: a Study Prospective, Randomized Placebo-controlled
Brief Title: Acute Influence of Resveratrol Supplementation and Beet Extract in Recovery After Exercise in Coronary Paths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luana Almeida Gonzaga, MD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UEPJMG
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Autonomic Nervous System Disease; Blood Pressure; Heart Rate
MeSH Terms: conditions — Coronary Artery Disease | interventions — Starch; Sucrose; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Protocol (Placebo Comparator): exercise and placebo capsules 500 mg (starch)
  Interventions: Other: Placebo Protocol
- Protocol Beet (Experimental): exercise and beet extract 500 mg
  Interventions: Other: Protocol Beet
- Protocol Resveratrol (Experimental): exercise and resveratrol capsules 500 mg
  Interventions: Other: Protocol Resveratrol
- Protocol Beet and Resveratrol (Experimental): exercise and beet extract 500mg and resveratrol capsules 500 mg
  Interventions: Other: Protocol Beet and Resveratrol

INTERVENTIONS:
Other: Placebo Protocol — ingestion of 500 mg of starch following 30 minutes of exercise (treadmill)
  Other Names: 500 mg of starch
  Arms: Placebo Protocol
Other: Protocol Beet — ingestion of 500 mg of beet extect following 30 minutes of exercise (treadmill)
  Other Names: 500 mg of beet extract
  Arms: Protocol Beet
Other: Protocol Resveratrol — ingestion of 500 mg of resveratrol following 30 minutes of exercise (treadmill)
  Other Names: 500 mg of resveratrol
  Arms: Protocol Resveratrol
Other: Protocol Beet and Resveratrol — ingestion 500 mg of beet extect and 500 mg of resveratrol following 30 minutes of exercise (treadmill)
  Other Names: 500 mg of beet extect and 500 mg of resveratrol
  Arms: Protocol Beet and Resveratrol

SUMMARY:
Introduction: Most cardiovascular diseases (CVD) can be prevented and controlled by adopting lifestyle changes, such as regular physical exercise and nutrition. Resveratrol and beverage extract promote beneficial health effects due to their nutritional properties. Objective: to analyze the effects of resveratrol supplementation and withdrawal extract on post-exercise recovery in coronary heart disease patients. Methods: men diagnosed with ischemic coronary artery disease will undergo four exercise protocols consisting of 30 minutes of aerobic exercise on an ergometric treadmill, with 5 minutes of warm-up, intensity of 30% of the heart rate reserve (HRR), followed by 25 minutes at intensity 60% of FCR and for a final 30 minutes of recovery in the supine position. Before each exercise protocol, all volunteers will consume: 500 mg of placebo (starch), or 500 mg of beetroot, or 500 mg of resveratrol and will also consume resveratrol and drink (500 mg each) 30 minutes before exercise. , the order of each supplementation will be done randomly. Cardiorespiratory parameters and heart rate variability (HRV) will be assessed at different times throughout the experimental procedure. To analyze the moments (rest versus recovery), the Bonferroni post-test will be used for parametric distribution or the Dunn post-test for non-parametric distribution. Statistical significance will be calculated at 5% for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* adult men over 45 years of age
* diagnosed with ischemic coronary artery disease and with preserved left ventricular function (above 50%), confirmed by a previous echocardiogram

Exclusion Criteria:

Volunteers who present at least one of the following characteristics will be excluded:

* smokers
* alcohol drinkers
* those who did not attend a cardiovascular rehabilitation program for at least 3 months prior to data collection
* individuals who have known infections, metabolic and respiratory diseases that could interfere in cardiac autonomic control, unstable angina, uncontrolled hypertension, significant valvular disease, uncontrolled metabolic disease (e.g., uncontrolled diabetes and thyroid disease)

Ages: 40 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | through study completion, an average of 1 hour
  Time and frequency domain of HRV

SECONDARY OUTCOMES:
Blood Pressure | through study completion, an average of 1 hour
  Systolic Blood Pressure and Diastolic Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual Paulista, Presidente Prudente, São Paulo, Brazil